CLINICAL TRIAL: NCT01270399
Title: Targeting ER-Golgi Homeostasis in an Advantageous Therapeutic Strategy in Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC10160-2010CTIL
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-03

CONDITIONS: The Combined Effect of Hsp90 Inhibitor and HDAC/Proteasome Inhibitors on Lung Cancer Cell Fate and ER-Golgi Homeostasis Will be Examined.

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- malignant neoplasm's cells
- natural cells

SUMMARY:
Lung cancer remains the most common cause of cancer-related death in the world. The major advances in treatment of lung cancer have brought only minor improvements in survival therefore novel systemic treatment methods are urgently needed.

Protein levels are regulated by the protein homeostasis network that generates and protects the protein fold (ER and Golgi included).

The heat shock protein 90 (Hsp90) is an essential molecular chaperon involved in the posttranslational folding and stability of proteins. Hsp90 inhibition leads to accumulation of unfolded proteins and ER stress. The therapeutic efficacy of such inhibition may be augmented by co-administering it with other drugs that disrupt ER-Golgi homeostasis like histone deacetylase (HDAC) or proteasome inhibitors. ER-Golgi homeostasis disruption affects a wide network of proteins and pathways as such affords a systemic target. Thus, the investigators aimed to examine the effect of combined treatment of Hsp90 antagonist with proteasome or HDAC inhibitors on human lung cancer cell lines and primary cells.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS WITH PROVED DIAGNOSIS OF LUNG CARCINOMA THAT ARE CANDIDATS FOR RADICAL SURGICAL TREATMENT

Exclusion Criteria:

* PATIENTS WITH SUSPICION FOR LUNG CARCINOMA WITHOUT PATHOLOGYCAL DIAFNOSIS BEFORE SURGERY

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: lung tissue with primary malignant neoplasm
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel